CLINICAL TRIAL: NCT03619785
Title: Ultrasound-guided (US) Serratus Anterior Plane Block (SAPB) for Acute Rib Fractures in the Emergency Department (ED)
Brief Title: US-guided SAPB for Rib Fractures in the ED
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Andrew A Herring (Other)
Collaborators: Oregon Health and Science University (Other); University of California, Los Angeles (Other)
Responsible Party: Sponsor-Investigator, Andrew A Herring, Associate Research Director, Department of Emergency Medicine, Highland Hospital, Alameda Health System
Organization: Alameda Health System (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 17-10102B
Record Dates: First submitted 2018-07-13; First posted 2018-08-08 (Actual); Last update posted 2018-12-19 (Actual); Status verified 2018-12

CONDITIONS: Rib Fractures; Rib Fracture Multiple
Keywords: Nerve Block; Serratus Anterior Plane Block; Ultrasound; Emergency Department
MeSH Terms: conditions — Rib Fractures; Emergencies | interventions — Bupivacaine; Fentanyl; Morphine; Hydromorphone; Hydrocodone; Acetaminophen; Ketorolac; Gabapentin; Ketamine; Ibuprofen

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Experimental (SAPB) (Experimental): Patients randomized to the experimental arm receive an ultrasound-guided serratus anterior plane block for their rib fracture pain.
  Interventions: Drug: Bupivacaine
- Control (Active Comparator): Patients randomized to the control arm receive usual pain control treatment in the emergency department.
  Interventions: Drug: Fentanyl, morphine, hydromorphone, hydrocodone, acetaminophen, ketorolac, gabapentin, ketamine, ibuprofen

INTERVENTIONS:
Drug: Bupivacaine — Patient will be positioned supine or in the lateral decubitus position on the side contralateral to the fracture(s). A 3.5 in 20-gauge needle, extension tubing, and a 30 mL syringe loaded with 0.25% bupivacaine and 3 mL of 1% lidocaine loaded in a 5 mL syringe with a 27-gauge needle will be prepared. The ribs, teres minor, latissimus dorsi, and serratus anterior will be identified with bedside US and the site of entry marked along the lateral aspect of the 4th-5th rib. The skin will be sterilized and lidocaine placed at the site of entry. The needle will be introduced at a steep angle and advanced in-plane, under US-guidance, to the plane superficial to the serratus anterior muscle. A test dose of normal saline will confirm proper needle tip placement with opening of the intramuscular layer. Injection with aliquots of 3-5 mL after negative aspiration will continue until 30mL of 0.25% bupivacaine are administered.
  Arms: Experimental (SAPB)
Drug: Fentanyl, morphine, hydromorphone, hydrocodone, acetaminophen, ketorolac, gabapentin, ketamine, ibuprofen — Oral or IV pain medication as needed.
  Arms: Control

SUMMARY:
The purpose of this randomized controlled study is to determine whether the serratus anterior plane block reduces pain more than the usual treatment for rib fractures in the same amount of time.

DETAILED DESCRIPTION:
Patients with unilateral rib fractures in the Highland Hospital Emergency Department who agree to participate will be randomized 1:1 to either the control group or the experimental group. Those in the control group will receive the usual oral and/or IV pain medication as needed. The experimental group will receive an ultrasound-guided serratus anterior plane block. Numerical pain rating scale scores at rest and when taking a deep breath will be recorded pre-intervention and at times 0, 20, 40, and 60. At time 60, patients who received the SAPB will receive sensory testing. Patients will be offered additional pain medication as needed at times 20, 40, and 60.

ELIGIBILITY:
Inclusion Criteria:

* Males and females 18 years and older, capable of providing informed consent indicating awareness of the investigational nature of the study, in keeping with institutional policy.
* Written informed consent must be obtained from each patient prior to entering the study.
* Patients with moderate to severe pain (NRS 4 to 10) as a result of one or more rib fractures occurring at levels T2-T8, measured on a self-reported NRS.

Exclusion Criteria:

* Patient refusal
* Patients with significant pain from other injuries (as determined at the discretion of the treating physician)
* Patients deemed critically ill by provider
* Patients with decompensated psychiatric disorders
* Pregnant patients (positive urine or serum B-HCG)
* History of heart block or bradycardia
* History of uncontrolled seizures
* Patients allergic to lidocaine, bupivacaine, ropivacaine, or morphine
* Patients with bilateral rib fractures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2018-11-06 (Actual); Primary Completion 2019-08-31 (Estimated); Study Completion 2019-08-31 (Estimated)

PRIMARY OUTCOMES:
Change in Numeric Pain Rating Scale score between time 0 and time 60 when comparing block and control groups | 60 minutes
  Change in Numeric Pain Rating Scale scores between time 0 and time 60 between block and control groups: Numeric Pain Rating Scale score at 0 minutes minus Numeric Pain Rating Scale score at 60 minutes, where a score of 0 is no pain and 10 is the worst pain the patient can imagine.

SECONDARY OUTCOMES:
Change in Numeric Pain Rating Scale score at rest versus when taking a deep breath when comparing block and control groups | 20, 40, 60 minutes
  Change in Numeric Pain Rating Scale score for resting chest pain and dynamic chest pain at 20, 40, and 60 minutes between block and control groups, where a score of 0 is no pain and 10 is the worst pain the patient can imagine.
Difference in total morphine equivalents | 1, 4, 12, and 24 hours
  Difference in total parenteral morphine equivalents received during study period (0 minutes to 60 minutes) and at 4, 12, and 24 hours (unless discharged from the hospital prior to 24 hours) in the block and control groups.
Successful analgesia for block group | 20, 40, 60 minutes
  Successful analgesia at 20, 40 and 60 minutes: Proportion of patients not receiving morphine dosing.
Non-opioid medications given (yes/no) | 20, 40, 60 minutes
  NSAID, APAP, Gabapentin administered in block versus control groups.
Adverse events | 60 minutes
  Proportion of patients with new onset of seizure, arrhythmias, hyper or hypotension (SBP<90 or >180), hypoxia, nausea, lightheadedness, vomiting.
Sensory testing | 60 minutes
  Sensory testing to cold stimulus (alcohol swab) in the block group along the lateral sternal, anterior axillary, and posterior axillary lines at the levels of T2-T10 using a 3-point scale: 0 (unchanged), 1 (reduced), or 2 (no sensation).

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Herring, MD, Principal Investigator — Alameda Health System - Highland Hospital; Josh Luftig, PA, Principal Investigator — Alameda Health System - Highland Hospital; Eben Clattenburg, MD, Principal Investigator — Alameda Health System - Highland Hospital; Daniel Mantuani, MD, MPH, Principal Investigator — Alameda Health System - Highland Hospital; Arun Nagdev, MD, Principal Investigator — Alameda Health System - Highland Hospital
Locations (1):
- Alameda Health System - Highland Hospital, Oakland, California, United States

IPD SHARING:
Plan to Share IPD: No